CLINICAL TRIAL: NCT05481034
Title: Simplified Meal Approach Study Using Hybrid Closed-loop Insulin Delivery in Youth and Young Adults With Type 1 Diabetes - a Randomised Controlled Two-centre Crossover Trial
Brief Title: Simplified Meal Approach Using Hybrid Closed-loop Insulin Delivery in Youth and Young Adults With Type 1 Diabetes
Acronym: SMASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lia Bally (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Prof. Dr.med. et Dr. phil., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SMASH
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Youth; Adolescents; Artificial pancreas system; Meal announcement
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified carbohydrate estimation first, exact carbohydrate estimation second (Experimental): In the first study period, participants will use the CamAPS FX system and adopt the "simplified meal announcement" (SMA) option to bolus for their meals. SMA comprises the selection of predefined carbohydrate quantities for meal insulin dosing. Meal carbohydrate contents will be set on an individual basis at the baseline visit. In the second study period, Participants will use the CamAPS FX system and insert the estimated grams of carbohydrates into the application as exactly as possible in order to bolus for their meals.
  Interventions: Device: SMA bolus option; Device: Exactly estimated carbohydrate content bolus option
- Exact carbohydrate estimation first, simplified carbohydrate estimation second. (Experimental): In the first study period, participants will use the CamAPS FX system and insert the estimated grams of carbohydrates into the application as exactly as possible in order to bolus for their meals. In the second study period, participants will use the CamAPS FX system and adopt the "simplified meal announcement" (SMA) option to bolus for their meals. SMA comprises the selection of predefined carbohydrate quantities for meal insulin dosing. Meal carbohydrate contents will be set on an individual basis at the baseline visit.
  Interventions: Device: SMA bolus option; Device: Exactly estimated carbohydrate content bolus option

INTERVENTIONS:
Device: SMA bolus option — SMA comprises the selection of predefined carbohydrate quantities for meal insulin dosing. Meal carbohydrate contents will be set on an individual basis at the baseline visit.
  Other Names: Simplified meal announcement bolus option
Device: Exactly estimated carbohydrate content bolus option — The carbohydrate content of meals is estimated in grams of carbohydrates prior to a meal bolus

SUMMARY:
The purpose of the study is to examine whether a simplified meal approach (as compared to exact carbohydrate counting) can alleviate the need of carbohydrate counting without worsening postprandial control in youth and young adults with type 1 diabetes using hybrid closed-loop insulin delivery with the Cambridge Artificial Pancreas FX System (CamAPS FX system).

DETAILED DESCRIPTION:
Optimal glycaemic control is the aim of diabetes care and critical in the prevention of diabetes-related complications. Despite advances in diabetes technologies and medications, many current youth and young adults (YYA) with type 1 diabetes (T1D) are not meeting desired glycaemic targets, representing a missed opportunity for improving lifetime outcomes.

A variety of factors including peer group influences, importance of body image, less parental oversight, greater risk-taking, and performance pressure challenge daily self-management in YYA with T1D. Disengagement from care and barriers for optimal glycaemic management in YYA have been mainly shown to be substantially influenced by perceived burden of daily tasks.

Although the recently introduced closed-loop systems, which link insulin delivery to sensor glucose levels, offer promising opportunities to improve glucose control in YYA with T1D, they still require the user to estimate carbohydrates. The perceived burden of exact carbohydrate counting (ECC), the limited evidence supporting its glycaemic benefit and corrective potential of algorithm-driven background insulin titration question its necessity during hybrid-closed loop insulin treatment. Instead, a simplified meal approach (SMA), which only requires the user to select the meal carbohydrate category (small/medium/large), has the potential to alleviate the burden of ECC during hybrid closed-loop insulin therapy whilst resulting in similar glycaemic benefits.

The investigators therefore hypothesize that a simplified meal approach (SMA) using the CamAPS FX system would achieve comparable glucose control compared with the use of the CamAPS FX system with ECC in YYA with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Type 1 diabetes as defined by the World Health Organization for at least 6 months
* Age between 12 and 20 years (inclusive)
* Proficient use of continuous glucose monitoring (CGM) or flash glucose monitoring (FGM) for at least 5 days in the past
* Glycated hemoglobin A1c (HbA1c) ≤12%
* The participant is willing to wear closed-loop devices
* The participant is willing to follow study specific instructions
* Negative urine-pregnancy test in sexually active female participants of childbearing potential at screening-visit

Exclusion Criteria:

* Any physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
* Known or suspected allergy against insulin
* Participant is pregnant or breast feeding or planning pregnancy within next 6.5 months
* Severe visual impairment
* Severe hearing impairment
* Lack of reliable telephone facility for contact
* Concomitant participation in another trial that interferes with the normal conduct of the study and interpretation of the study results
* Participant not proficient in German

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Percentage of time with sensor glucose measurements between 3.9 and 10.0 mmol/L | From the first day of the respective study period to 3 months thereafter
  The percentage of time with sensor glucose measurements between 3.9 and 10.0 mmol/L will be compared between both intervention arms. Primary analysis will be carried out according to a non-inferiority framework.

SECONDARY OUTCOMES:
Time spent with sensor glucose values above target (>10.0 mmol/L) | From the first day of the respective study period to 3 months thereafter
  Percentage of time spent with sensor glucose values above target (>10.0 mmol/L)
Time spent with sensor glucose values >13.9 mmol/L (%) | From the first day of the respective study period to 3 months thereafter
  Percentage of time spent with sensor glucose values >13.9 mmol/L (%)
Time spent with sensor glucose measurements < 3.9 mmol/L | From the first day of the respective study period to 3 months thereafter
  The percentage of time with sensor glucose measurements < 3.9 mmol/L (%)
Time spent with sensor glucose measurements < 3.0 mmol/L | From the first day of the respective study period to 3 months thereafter
  The percentage of time with sensor glucose measurements < 3.0 mmol/L (%)
Time spent with sensor glucose measurements between < 3.9 mmol/L and 7.8 mmol/L (%) | From the first day of the respective study period to 3 months thereafter
  The percentage of time with sensor glucose between < 3.9 mmol/L and 7.8 mmol/L (%)
Mean sensor glucose level (mmol/L) | From the first day of the respective study period to 3 months thereafter
  Mean of all sensor glucose levels (mmol/L)
HbA1c | At baseline and at the predefined study visits (3 months after the start of the respective periods)
  Glycated hemoglobin A1c (%)
Mean peak postprandial glucose | From the first day of the respective study period to 3 months thereafter
  Mean peak postprandial glucose (mmol/L) assessed within 180min following main meals (defined as carbohydrate amounts >25g entered into the CamAPS app by the participants).
Coefficient of sensor glucose variation (%) | From the first day of the respective study period to 3 months thereafter
  Coefficient of sensor glucose variation (%)
Standard deviation of sensor glucose variation (mmol/L) | From the first day of the respective study period to 3 months thereafter
  Standard deviation of sensor glucose variation (mmol/L)
Glucose Management Indicator (%) | From the first day of the respective study period to 3 months thereafter
  Glucose Management Indicator (%)
Number of clinically significant hypoglycaemia (number of events with sensor glucose <3.9 mmol/L for at least 15min) | From the first day of the respective study period to 3 months thereafter
  Number of events with sensor glucose <3.9 mmol/L for at least 15min
Extended hypoglycaemia event rate (number of events with sensor glucose <3.9 mmol/L lasting at least 120min) | From the first day of the respective study period to 3 months thereafter
  Number of events with sensor glucose <3.9 mmol/L lasting at least 120min
Extended hyperglycaemia event rate (number of events with sensor glucose >13.9 mmol/L lasting at least 120min) | From the first day of the respective study period to 3 months thereafter
  Number of events with sensor glucose >13.9 mmol/L lasting at least 120min
Proportion of participants with sensor glucose in the target range (3.9 - 10.0 mmol/L for >70% of the time. | From the first day of the respective study period to 3 months thereafter
  Proportion of participants with sensor glucose in the target range (3.9 - 10.0 mmol/L for >70% of the time.

OTHER OUTCOMES:
Total daily basal insulin dose | From the first day of the respective study period to 3 months thereafter
  Mean total daily basal insulin dose infused
Total daily bolus insulin dose | From the first day of the respective study period to 3 months thereafter
  Mean total daily bolus insulin dose infused
Percentage of time of closed-loop operation including engagement with specific functionalities | From the first day of the respective study period to 3 months thereafter
  Utility evaluation
Diabetes Distress Scale | At the predefined study visit 3 months after the start of the respective period.
  Measurement of distress associated with the use of closed-loop insulin delivery using the Diabetes Distress questionnaire
Hypoglycaemia confidence scale | At the predefined study visit 3 months after the start of the respective period.
  HCS is a 9-item self-report scale that examines the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems
Psychosocial factors important to quality of life | At the predefined study visit 3 months after the start of the respective period.
  These factors include anxiety, stress, depressions, etc.
Food Frequency Questionnaire to assess dietary intake habits | At the predefined study visit 3 months after the start of the respective period.
  Dietary intake (quantity and quality)
Number of severe hypoglycaemia events | From the first day of the respective study period to 3 months thereafter
  Hypoglycaemia requiring third-party assistance to administer carbohydrates or other resuscitative action
Diabetic ketoacidosis | From the first day of the respective study period to 3 months thereafter
  ADA definition
Significant ketonaemia | From the first day of the respective study period to 3 months thereafter
  Value > 3.0 mmol/L
Nature and severity of adverse events | From the first day of the respective study period to 3 months thereafter
  AE including SADE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD PhD, Principal Investigator — University hospital of Bern
Locations (2):
- Switzerland (2):
  - Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital and University of Bern, Bern, Switzerland, Bern
  - Department of Paediatric Endocrinology and Diabetes, University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data will be shared after inquiry via a validated sharing platform (yet to be defined). Anonymised data packages will be available once the final study results are published in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the study results in a peer-reviewed journal.
Access Criteria: Contact with and approval by the corresponding author

REFERENCES:
- [Derived] Laesser CI, Piazza C, Schorno N, Nick F, Kastrati L, Zueger T, Barnard-Kelly K, Wilinska ME, Nakas CT, Hovorka R, Herzig D, Konrad D, Bally L. Simplified meal announcement study (SMASH) using hybrid closed-loop insulin delivery in youth and young adults with type 1 diabetes: a randomised controlled two-centre crossover trial. Diabetologia. 2025 Feb;68(2):295-307. doi: 10.1007/s00125-024-06319-w. Epub 2024 Nov 19. PMID 39560745